CLINICAL TRIAL: NCT02961465
Title: Effectiveness and Safety of Sacral Neuromodulation in Patients With Idiopathic Slow-transit Constipation Refractory to Conservative Treatments
Brief Title: Effectiveness and Safety of Sacral Neuromodulation in Patients With Idiopathic Slow-transit Constipation
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch National Health Care Institute (Other); Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: METC161044
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Constipation; Surgery
Keywords: Sacral neuromodulation; Constipation; Slow-transit constipation; Surgery; Colorectal surgery; Cost-effectiveness; Quality of life
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sacral Neuromodulation (SNM)
  Interventions: Device: Sacral Neuromodulation

INTERVENTIONS:
Device: Sacral Neuromodulation — SNM starts with a screening phase. In this phase a tined lead is inserted into the third sacral foramen and attached to an external stimulator, after which the patient enters a four-week stimulation test period.
  If the screening phase is successful (defecation frequency (DF) ≥3 a week), the external stimulator is changed for a pacemaker that is implanted in the buttocks. If the screening phase is unsuccessful (DF <3 a week), the lead is explanted. Patients are asked to limit the use of additional conservative treatments for constipation (such as laxatives and colonic irrigation) to what is necessary to relieve (the most severe) complaints. What is necessary to relieve complaints is determined by the patient.
  Other Names: Medtronic Interstim Therapy System

SUMMARY:
Rationale: Previous reviews showed that the evidence regarding the effectiveness of sacral neuromodulation (SNM) in patients with therapy-resistant, idiopathic (slow-transit) constipation is of suboptimal quality. Furthermore, there is no estimate of costs and cost-effectiveness in this patient group.

Study design: A prospective cohort study with one group. This study is conducted next to a randomized controlled clinical trial (RCT) on 'the effectiveness and cost-effectiveness of sacral neuromodulation in patients with idiopathic slow-transit constipation refractory to conservative treatments' (for more information ClinicalTrial.gov ID: NCT02961582). This RCT is part of a temporary reimbursement arrangement, called conditional reimbursement of health care (in Dutch: Voorwaardelijke Toelating) of the National Health Care Institute (Zorginstituut Nederland). As part of this arrangement, the Ministry of Health, Welfare and Sports requires that SNM remains available for eligible patients during the conditional reimbursement period, also when inclusion of the RCT has ended. Furthermore, the Ministry requires that patients who received personalized conservative treatment in the RCT (control group), are offered SNM after completion of their follow-up of 6 months. As a result, the National Health Care Institute requires that the patients who receive SNM outside the RCT are included in a prospective cohort study to be able to collect data on them.

Aim: The aim of this prospective cohort study is to collect more (but uncontrolled) information regarding the safety and effectiveness of SNM.

Study population: Adolescent (14-17 years) and adult (18-80 years) patients with idiopathic slow-transit constipation refractory to conservative treatment.

Intervention: The intervention is SNM, a minimally invasive surgical procedure consisting of two phases. In the screening phase an electrode is inserted near the third sacral nerve and connected to an external stimulator. If the screening phase is successful (average defecation frequency (DF) ≥3 a week), the electrode is connected to a pacemaker that is implanted in the buttocks of the patient. If not successful, the pacemaker will be removed and patients receive conservative treatment.

Main study parameters/endpoints: The primary outcome is treatment success at 6 months, defined as an average DF of ≥3 a week according to a 3-week defecation diary and safety. Secondary outcomes are straining, sense of incomplete evacuation, constipation severity and generic (health-related) quality of life ((HR)QOL).

ELIGIBILITY:
Inclusion Criteria:

* An average defecation frequency (DF) of <3 per week based on a 3-week defecation diary (patient-reported)
* Meet at least one other criterion of the Rome-IV criteria for idiopathic constipation based on the 3-week defecation diary (1)
* Refractory to conservative treatment
* Age: 14-80 years
* Slow-transit constipation

  (1) Rome-IV criteria for idiopathic constipation:
* Straining during ≥25% of defecations
* Lumpy or hard stools in ≥25% of defecations
* Sensation of incomplete evacuation for ≥25% of defecations
* Sensation of anorectal obstruction/blockage for ≥25% of defecations
* Manual manoeuvres to facilitate ≥25% of defecations

Exclusion Criteria:

* Obstructed outlet syndrome (objectified by defeacography)
* Irritable bowel syndrome (Rome-IV criteria for irritable bowel syndrome)
* Congenital or organic bowel pathology
* Rectal prolapse
* Anatomical limitations preventing placement of an electrode
* Skin and perineal disease with risk of infection
* Previous large bowel/rectal surgery
* Stoma
* Coexisting neurological disease
* Significant psychological co-morbidity as assessed subjectively by the investigator
* Being or attempting to become pregnant during study follow-up

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adolescents (14-17 years) and adults (18-80 years) with idiopathic slow-transit constipation refractory to conservative treatment. As data regarding this population is limited it is virtually impossible to provide precise numbers of this patient population. However, some numbers are known:
  * Average prevalences of idiopathic constipation of 16% and 19.2% are reported in Europe
  * Of all patients treated for constipation, 5.6% is treated at the hospital
  * It is estimated that 1% of the constipation patients who are treated with conservative treatment in hospitals, are unresponsive and are eligible for sacral neuromodulation
  * Over the last 6 years, annually, on average, 25 patients were treated with SNM at the Maastricht UMC+ and the Groene Hart Ziekenhuis Gouda
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment success at 6 months | 6 months
  Treatment success is defined as an average defecation frequency of ≥ 3 a week based on a patient-reported defecation diary over a period of 3 weeks
Complications/adverse events | 6 months
  Reported by the clinician in a case report form (CRF)

SECONDARY OUTCOMES:
Proportion of patients with a 50% reduction in the proportion of defecations with straining | Baseline, 1, 3 and 6 months, (12 months)
  The proportion of defecations with straining is derived from the data in the 3 week defecation diary. The reported proportion of defecations with straining is compared with the proportion of defecations with straining at baseline. Patients are divided in two groups: 1) ≥50% reduction in the proportion of defecations with straining and 2) <50% reduction in the proportion of defecations with straining. In patients who still have the pacemaker at 6 months, outcomes are als measured 12 months after inclusion to monitor the longer term effectiveness and safety of SNM.
Proportion of patients with a 50% reduction in the proportion of defecations with a sense of incomplete evacuation | Baseline, 1, 3 and 6 months, (12 months)
  The proportion of defecations with a sense of incomplete evacuation is derived from the data in the 3 week defecation diary. The reported proportion of defecations with a sense of incomplete evacuation is compared with the proportion of defecations with a sense of incomplete evacuation at baseline. Patients are divided in two groups: 1) ≥50% reduction in the proportion of defecations with a sense of incomplete evacuation and 2) <50% reduction in the proportion of defecations with a sense of incomplete evacuation. In patients who still have the pacemaker at 6 months, outcomes are als measured 12 months after inclusion to monitor the longer term effectiveness and safety of SNM.
Constipation severity | Baseline, 1, 3 and 6 months, (12 months)
  Displayed with the score from the Wexner constipation score (WCS). In patients who still have the pacemaker at 6 months, outcomes are als measured 12 months after inclusion to monitor the longer term effectiveness and safety of SNM.
Generic (HR)QOL | Baseline, 1, 3 and 6 months, (12 months)
  Displayed with the score from the EQ-5D-5L. In patients who still have the pacemaker at 6 months, outcomes are als measured 12 months after inclusion to monitor the longer term effectiveness and safety of SNM.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie O Breukink, Dr., Principal Investigator — Maastricht University Medical Centre; Carmen D Dirksen, Prof. dr., Principal Investigator — Maastricht University Medical Centre
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Groene Hart Ziekenhuis, Gouda, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mugie SM, Benninga MA, Di Lorenzo C. Epidemiology of constipation in children and adults: a systematic review. Best Pract Res Clin Gastroenterol. 2011 Feb;25(1):3-18. doi: 10.1016/j.bpg.2010.12.010. PMID 21382575
- [Background] Suares NC, Ford AC. Prevalence of, and risk factors for, chronic idiopathic constipation in the community: systematic review and meta-analysis. Am J Gastroenterol. 2011 Sep;106(9):1582-91; quiz 1581, 1592. doi: 10.1038/ajg.2011.164. Epub 2011 May 24. PMID 21606976
- [Background] van Wunnik BP, Peeters B, Govaert B, Nieman FH, Benninga MA, Baeten CG. Sacral neuromodulation therapy: a promising treatment for adolescents with refractory functional constipation. Dis Colon Rectum. 2012 Mar;55(3):278-85. doi: 10.1097/DCR.0b013e3182405c61. PMID 22469794